CLINICAL TRIAL: NCT04918914
Title: Off Label Use of Dapsone in SARS-CoV-2 Hospitalized Patients
Brief Title: Critical Care Results of SARS-CoV-2 ARDS by Dapsone and Standard COVID-19 Treatment
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunt Regional Medical Center (Other)
Responsible Party: Principal Investigator, Badar Kanwar, Principal Investigator, Hunt Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Badar Kanwar
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2; Hypoxia; ARDS
MeSH Terms: conditions — Hypoxia | interventions — Dapsone

STUDY DESIGN:
Intervention Model Description: Addition of dapsone to COVID19 patient treated with standard treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Other)
  Interventions: Drug: Dapsone 100 MG

INTERVENTIONS:
Drug: Dapsone 100 MG — Dapsone 100-200 md orally daily, along with Cimetadine 400 mg PO TID

SUMMARY:
Abstract Background: Clinicians in pulmonary critical care medicine and critical care medicine considered dapsone administration to treat SARS-CoV-2 inflammasome. Dapsone is useful in the molecular regulation of Nod-like receptor family pyrin domain-containing 3 (NLRP3).

Objective: To study the targeting of NLRP3 itself or up-/downstream factors of the NLRP3 inflammasome by dapsone must be responsible for its observed preventive effects, functioning as a competitor.

Methods:

Patients who were on standard COVID-19 therapy are also after obtaining off label uses and explanation of side effects are started on dapsone 100-200 mg daily along with Cimetadine 400 mg three times daily.

DETAILED DESCRIPTION:
We are investigating in prospective ongoing non-randomized case study effects of addition of dapsone 100-200 mg daily in addition to standardized recommended treatment versus a a cohort of patient admitted at our institution since October 2020 versus a group that only received standardized treatment. Our primary out comes are decrease in FIO2 requirement leading to discharge from hospital and decrease in over all mortality between group treated with only standardized recommended treat versus group with addition of dapsone and cimetadine.

An objective criteria of improvement, was used for effectiveness of therapy.

A. a reduction in the FIO2 requirement and

B. a decrease in the progression of hypoxia. We treated the patients with standard COVID-19 ARDS treatment with dapsone 100 mg to target NLRP3 inflammasomes.

ELIGIBILITY:
Inclusion Criteria:

1. All, PCR confirmed cases of COVID-19

Exclusion Criteria:

1. Only consenting consenting patients

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Critical Care Results of SARS-CoV-2 ARDS by Dapsone and Standard COVID-19 Treatment | 1 year
  1. Decrease in overall mortality between groups treated with standardized recommended composite therapy for COVID-19 versus group of Standardized therapy plus addition of dapson and cimedatine

CONTACTS AND LOCATIONS:
Locations (1):
- Hunt Regional Medical Center, Greenville, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code